CLINICAL TRIAL: NCT05399186
Title: Incidence of Modifiable Risk Factors and Their Association With Infections in Primary Elective Arthroplastic Surgery
Brief Title: Arthroplasty and Modifiable Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Sigurbergur Karason, Professor, Landspitali University Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20220508
Record Dates: First submitted 2022-05-19; First posted 2022-06-01 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Total Joint Arthroplasty; Risk Reduction; Surgical Site Infection; Prosthetic-joint Infection; Postoperative Complications
MeSH Terms: conditions — Risk Reduction Behavior; Surgical Wound Infection; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: A prospective non-randomized quality control study before and after an intervention regarding preoperative preparation for total joint arthroplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual care group - receiving traditional preoperative preparation and assessment (1 week) prior to total joint arthroplastic surgery
- Early preoperative assessment and optimization (Experimental): Interventional group - receiving early preoperative assessment and optimization (6-12 months) in wait of total joint arthroplastic surgery
  Interventions: Other: Early preoperative assessment and optimization

INTERVENTIONS:
Other: Early preoperative assessment and optimization — The interventional group received early preoperative assessment and optimization (6-12 months) prior to total joint arthroplastic surgery in cooperation between hospital and primary care
  Arms: Early preoperative assessment and optimization

SUMMARY:
Hip and knee total joint arthroplasty are one of the most frequently performed surgery worldwide. However, prosthetic joint infection remains a devastating complication of them, associated with severe morbidity, increased mortality and huge costs. Several underlying medical conditions that have been identified as independent risk factors for development of prosthetic joint infection.

The hypothesis of the study is that by utilizing the waiting time for operation (6 -12 months) to improve the state of known modifiable risk factors the frequency of prosthetic joint infection may be decreased. This optimization was established with co-operation between hospital and primary care.

Therefore a prospective non-randomized quality control study before and after an intervention regarding preoperative preparation for total joint arthroplasty of either hip or knee was planned.

The control arm was included one week prior to surgery at the anesthesia preoperative assessment outpatient clinic and were operated on between 27/8 2018 and 7/9 2020 and consists of 738 patients.

Inclusion of the interventional arm happened at the orthopedic outpatient clinic from 2/1 2019 - 30/1 2021, 6 -12 months prior to surgery and an appointment with their general physician ensured within 3 weeks for further evaluation. Enlisted have been 1010 patients, operation of them started 25/3 2019 and to date 710 patients have been operated on, but due to delays caused by Covid-19 (SARS-CoV-2) surgery of them is still ongoing.

The effect of the intervention will be evaluated with by comparison of patient characteristics and frequency of surgical site and prosthetic joint infections before and after.

DETAILED DESCRIPTION:
Hip and knee total joint arthroplasty allow effective treatment of disability and pain due to joint destruction, and are one of the most frequently performed surgery worldwide. Surgical-site infections remain a serious complication of total joint arthroplasty, occurring in 1-7% of cases. The most severe form of surgical site infection, prosthetic joint infection is a devastating complication associated with severe morbidity, increased mortality and huge costs. There are several underlying medical conditions that have been identified as independent risk factors for development of prosthetic joint infection that might be improved before operation, called modifiable risk factors, namely pre-operative anemia, obesity, diabetes, poor nutritional status, smoking and physical activity.

The hypothesis of the study is that by utilizing the waiting time for operation (6 -12 months) to improve the state of known modifiable risk factors the frequency of prosthetic joint infection may be decreased. This optimization was established with co-operation between hospital and primary care.

Therefore a prospective non-randomized quality control study before and after an intervention regarding preoperative preparation for total joint arthroplasty of either hip or knee, comparing patient characteristics and outcome was planned.

Control Arm: Inclusion of 'usual care' patients started 20/8 2018 one week prior to surgery at the anesthesia preoperative assessment outpatient clinic. At that point in time there were 561 patients already on a waiting list for either hip or knee arthroplastic surgery. The next four months to 31/12 2018 66 more patients were added to the study. After 1/1 2019 (when collection to the interventional part had started) further 111 patients were added (15% of the 'usual care' group). These were patients where it had been missed to offer or had declined participation in the interventional arm of the study at the orthopedic outpatient clinic and when discovered at the preoperative clinic one week prior to surgery were offered participation in the 'usual care' arm as they had received traditional preoperative preparation. Operation of these patients started at 27/8 2018 and lasted to 7/9 2020 and consists of total of 738 individuals.

Interventional arm: Inclusion into the interventional arm of the study occurred between 2/1 2019 to 30/1 2021, 6 -12 months prior to surgery at the orthopedic outpatient clinic, ensuring an appointment with the patient general physician within 3 weeks afterwards to further analyze results of blood test and assess if further tests, treatments or consultation of other specialists would be preferred to optimize their condition. Patients at extremes of BMI also had a nutritional advice at the hospital. Enlisted have been 1010 patients, operation of them started 25/3 2019 and to date 710 patients have been operated on, but due to delays caused by COVID-19 (SARS-CoV-2) surgery of them is still ongoing.

Outcome variables: Information was gathered regarding age, gender, smoking, comorbidities, type of surgery, type of anesthesia, ASA classification, weight, physical activity, laboratory values (Hb, Glu, HbA1c, Albumin. Lymphocytes, D-vitamin), blood transfusions and length of stay. Postoperative follow up happened first 3 weeks postoperatively at primary care for suture removal and then 6 weeks at the outpatient orthopedic clinic. Notes from these visits were studied to identify surgical site complications, including surgical site infection, prosthetic joint infection, surgical site drainage, bleeding, dehiscence, and hematoma and evaluated according to CDC's National Healthcare Safety Network and PJI diagnosis. Also, a two year follow will occur by analysis of patient journal in regards of complications of the arthroplasty.

Statistical methods. Patient demographics will be described as median (interquartile range) for continuous variables, and number (percentage) for categorical variables. Mean and standard deviation (SD) will be reported for normally distributed data. A univariate association between the presence of modifiable risk factors and the presence of postoperative surgical site infection will be assessed using chi-squared test for categorical variables and t-test for continuous variables. As this is a descriptive study and incidence of modifiable risk factors not known in the cohort no assessment of power was performed prior to analysis. To study if there is a difference between the groups a t-test or non-parametric Wilcoxon rank sum test or Hotelling's t will be used for continuous parameters, and chi-squared test or Fisher's exact test to compare categorical parameters. Poisson regression or negative binominal regression of zero inflated regression will be used to study if a difference in the frequency of complications has occurred after the intervention. These methods might be subjected to change if unexpected factors arise during analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing elective primary arthroplasty of either hip or knee at Landspitali University Hospital

Exclusion Criteria:

* Contraindications for operation detected after inclusion. Patients having an operation on another joint within the inclusion period were not re-included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1484 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Surgical site infection | 6 weeks postoperatively
  Evaluated according to CDC's National Healthcare Safety Network
Number of Participants with Surgical site infection | 2 years postoperatively
  Evaluated according to CDC's National Healthcare Safety Network
Number of Participants with Prosthetic joint infection | 6 weeks postoperatively
  Evaluated according to CDC's National Healthcare Safety Network
Number of Participants with Prosthetic joint infection | 2 years postoperatively
  Evaluated according to CDC's National Healthcare Safety Network

SECONDARY OUTCOMES:
Preoperative anemia according to WHO's definition | At inclusion, 1 week prior to and one day after surgery
  Hemoglobin in blood - Preoperative anemia was defined according to WHO's definition as a haemoglobin concentration of <120 g/l and < 130 g/l in women and men, respectively, and divided into mild (110 - 120/130 g/L per gender), moderate (80-109 g/L) and severe (<80 g/L).
Control of diabetes | At inclusion, 1 week prior to and one day after surgery
  HbA1c level - Patients were considered to have diabetes if they had received this diagnosis preoperatively or had a HbA1c level >47 mmol/mol. Non-diabetic patients were considered to have dysglycemia if HbA1c was 42 - 47 mmol/mol and undiagnosed diabetes if HbA1c >47mmol/mol.
Indication of poor glucose control | At inclusion, 1 week prior to and one day after surgery
  Serum Glucose level
Nutritional status | At inclusion, 1 week prior to and one day after surgery
  S- albumin - Patients with <35g/L (3.5 g/dL) were considered to be at risk of malnutrition
Nutritional status | At inclusion, 1 week prior to and one day after surgery
  Lymphocyte count - Patients with <1,5 x 10E9/L 32 were considered to be at risk of malnutrition
Nutritional status | At inclusion, 1 week prior to and one day after surgery
  D-Vitamin - Patients with 25OHD concentration < 50 nmol/L were defined as having a deficiency
Smoking | At inclusion, 1 week prior to surgery
  Information of smoking habits were acquired through a questionnaire and divided into those that had quit smoking more than a year ago >than 6 months ago, >6 weeks ago, less than 6 weeks ago and current smokers
Physical activity | At inclusion, 1 week prior to surgery
  Information of amount of weekly physical activity was acquired through a questionnaire and divided into two classes, zero to two times per week and three to five times per week. Each occasion was graded from 1 to more than 60 minutes.
Other postoperative complications | up to two years postoperatively
  Information from health records

CONTACTS AND LOCATIONS:
Overall Officials: Sigurbergur Karason, Professor, Principal Investigator — Landspitali University Hospital
Locations (1):
- Landspitali University Hsopital, Reykjavik, Hringbraut, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and 10 years afterwards
Access Criteria: Upon reasonable request